CLINICAL TRIAL: NCT03861520
Title: Correlation Between Ultrasonographic Fetal Soft Markers and Aneuploidy
Brief Title: Ultrasonographic Fetal Soft Markers and Aneuploidy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Ahmed Bassiouny, Assistant Professor, Cairo University
Other Study IDs: 12019
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Soft Markers
Keywords: Anomaly scan; Anuploidy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fetal karyotyping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 16-24 weeks Pregnant womes: Pregnant Women at (16-24) weeks of gestation for mid trimester anomaly scan with one sonographic fetal soft marker or more.
  Interventions: Device: Midtrimester anomaly scan; Genetic: Fetal Karyotyping

INTERVENTIONS:
Device: Midtrimester anomaly scan — A detailed anomaly scan to detect soft markers at 16 to 24 weeks pregnancy
  Other Names: 2nd trimester anomaly scan
Genetic: Fetal Karyotyping — Fetal karyotyping after birth to confirm chromosomal anomaly diagnosed clinically

SUMMARY:
The purpose of this study is to investigate the prevalence of soft markers which will be identified during a second trimester ultrasound. Secondary aims were to estimate the association between the soft markers and trisomies 13, 18 and 21 as well as the effect on the number of invasive tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant woman between (16-24) weeks of gestation.
2. singelton pregnancy.

Exclusion Criteria:

1. Multiple pregnancies.
2. Mental condition rendering the patients unable to understand the nature and scope of the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women at (16-24) weeks of gestation for mid trimester anomaly scan with one sonographic fetal soft marker or more
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
To study the association between soft markers identified at second trimester ultrasound and aneuploidy. | 1 year
  fetal soft markers detection which include the following:
  * choroid plexus cyst.
  * Mild ventriculomegaly.
  * Enlarged cistern magna.
  * Nasal bone hypoplasia.
  * Increased nuchal fold.
  * Echogenic cardiac focus.
  * Single umbilical artery.
  * Pyelectasis.
  * Echogenic bowl.
  * Short femur.
  * Short humerus.
  All data will be collected and statistics will be done for the correlation between one or more soft markers with structural anomalies and its relation with aneuploidy.

CONTACTS AND LOCATIONS:
Overall Officials: Maha M Mossad, MD, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No